CLINICAL TRIAL: NCT05013554
Title: A Phase 1/1b Open-label, First-in-human, Single Agent, Dose Escalation and Expansion Study for the Evaluation of Safety, Pharmacokinetics, Pharmacodynamics, and Anti-tumor Activity of SAR443216 in Participants With Relapsed/Refractory HER2 Expressing Solid Tumors.
Brief Title: Dose Escalation and Expansion Study of SAR443216 in Participants With Relapsed/Refractory HER2 Expressing Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TED16925; U1111-1253-2233 (Registry Identifier: ICTRP); 2023-506852-26-00 (Registry Identifier: CTIS); 2021-000086-32 (EudraCT Number)
Record Dates: First submitted 2021-08-12; First posted 2021-08-19 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Neoplasm Malignant; Breast Cancer; Lung Neoplasm Malignant; Gastric Cancer; Neoplasm
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Lung Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- SAR443216-Dose Escalation (Experimental): Participants with metastatic solid tumors that express HER2 in tumor tissue and/or with HER2 aberration will receive SAR443216 as intravenous (IV) infusion or subcutaneous (SC) injection.
  Interventions: Drug: SAR443216 IV; Drug: SAR443216 SC
- SAR443216-Dose Expansion - metastatic breast cancers with HER2 high expression: Cohort A (Experimental): Participants with metastatic breast cancers with HER2 high expression (with amplification) will receive SAR443216 as intravenous (IV) infusion.
  Interventions: Drug: SAR443216 IV
- SAR443216-Dose Expansion- metastatic breast cancers with HER2 low expression: Cohort B (Experimental): Participants with metastatic breast cancers with HER2 low expression or HER2 mutation (without amplification) will receive SAR443216 as intravenous (IV) infusion.
  Interventions: Drug: SAR443216 IV
- SAR443216-Dose Expansion- metastatic gastric cancers with HER2 low expression: Cohort C (Experimental): Participants with metastatic gastric cancers with HER2 low expression or HER2 mutation (without amplification) will receive SAR443216 as intravenous (IV) infusion.
  Interventions: Drug: SAR443216 IV
- SAR443216-Dose Expansion - metastatic NSCLC with HER2 low or high expression: Cohort D (Experimental): Participants with metastatic NSCLC with HER2 low or high expression and/or HER2 mutation will receive SAR443216 as intravenous (IV) infusion.
  Interventions: Drug: SAR443216 IV

INTERVENTIONS:
Drug: SAR443216 IV — Pharmaceutical form: Powder for solution; Route of administration: IV infusion
Drug: SAR443216 SC — Pharmaceutical form: Powder for solution; Route of administration: SC injection
  Arms: SAR443216-Dose Escalation

SUMMARY:
Primary Objectives:

Part 1 (Dose Escalation)

* To determine the MTD/maximum administered dose (MAD) of SAR443216 administered as a single agent in participants with HER2 expressing solid tumors and determine the RD(s) for intravenous (IV) and subcutaneous (SC) administration in the dose escalation part.
* To determine the safety of SAR443216 after intravenous (IV) and subcutaneous (SC) administration.

Part 2 (Dose expansion)

• To assess preliminary clinical activity of single agent SAR443216 at the RD(s) in participants with HER2 expressing solid tumors, with various levels of HER2 expression.

Secondary Objectives:

Part 1 • To assess preliminary clinical activity of single agent SAR443216 after IV and SC administration at the RD(s) in participants with HER2 expressing solid tumors, with various levels of HER2 expression.

Part 2

• To determine the safety of SAR443216.

Part 1 and 2

* To characterize the pharmacokinetic (PK) profile of SAR443216 when administered as a single agent after IV and SC (Part 1 only) administration.
* To evaluate the immunogenicity of SAR443216 after IV and SC administration.
* To assess preliminary clinical activity of single agent SAR443216 at the RD(s) in participants with HER2 expressing solid tumors, with various levels of HER2 expression.

DETAILED DESCRIPTION:
The expected duration of study intervention for participants may vary, based on progression date; median expected duration of study per participant is estimated to be:

* 7.5 months (up to 1 month for screening, a median of 3.5 months for treatment, and a median of 3 months for long term follow-up) in escalation.
* 9.5 months (up to 1 month for screening, a median of 5.5 months for treatment, and a median of 3 months for long term follow-up) in expansion.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be ≥ 18 years of age
* Histologically or cytologically confirmed diagnosis of metastatic solid tumors
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* All participants should have at least 1 measurable disease per RECIST v1.1. An irradiated lesion can be considered measurable only if progression has been demonstrated on the irradiated lesion.
* Body weight within [45 - 150 kg] (inclusive)
* All Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Capable of giving signed informed consent

Exclusion Criteria:

* Any clinically significant cardiac disease
* History of or current interstitial lung disease or pneumonitis
* Uncontrolled or unresolved acute renal failure
* Prior solid organ or hematologic transplant.
* Known positivity with human immunodeficiency virus (HIV), known active hepatitis A, B, and C, or uncontrolled chronic or ongoing infectious requiring parenteral treatment.
* Receipt of a live-virus vaccination within 28 days of planned treatment start
* Participation in a concurrent clinical study in the treatment period.
* Inadequate hematologic, hepatic and renal function
* Participant not suitable for participation, whatever the reason, as judged by the Investigator, including medical or clinical conditions.

The above information is not intended to contain all considerations relevant to the potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Part 1: Dose Escalation Determine the MTD/maximum administered dose (MAD) and RD(s) of SAR443216 | Cycle 1, cycle duration is 28 days for 2-week lead-in schedule and 35 days for 3-week lead-in schedule
  Incidence of study dose limiting toxicities (DLTs)
Part 1: Dose Escalation: Safety of SAR443216 | Baseline until end of study, up to approximately 7.5 months
  Incidence of treatment emergent adverse events (TEAEs), serious adverse events (SAEs), and lab abnormalities according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
Part 2: Dose Expansion Objective response rate (ORR) of SAR443216 in all participants | From date of enrollment until the end of treatment, up to approximately 5.5 months
  Objective response rate is defined as the proportion of participants who achieve a complete response (CR) or partial response (PR) per RECIST v1.1.
Part 2: Dose Expansion Duration of response (DoR) of SAR443216 in all participants. | From date of enrollment until the end of treatment, up to approximately 5.5 months
  Duration of response per RECIST v1.1 is defined as the interval from the first documentation of CR or PR to the earlier of the first documentation of definitive disease progression or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Part 1: Objective response rate (ORR) of SAR443216 in all participants | From date of enrollment until the end of treatment, up to approximately 3.5 months
  Objective response rate is defined as the proportion of participants who achieve a complete response (CR) or partial response (PR) per RECIST v1.1.
Part 1: Duration of response (DoR) of SAR443216 in all participants | From date of enrollment until the end of treatment, up to approximately 3.5 months
  Duration of response per RECIST v1.1 is defined as the interval from the first documentation of CR or PR to the earlier of the first documentation of definitive disease progression or death due to any cause, whichever occurs first
Part 1 and Part 2: Progression Free Survival (PFS) | From date of enrollment until the end of treatment, up to approximately 3.5 months for Part1 and 5.5 months for Part 2
  Progression free survival (PFS) will be assessed by the Investigator per RECIST v1.1 and will be summarized using the Kaplan-Meier method
Part 2: Safety of SAR443216 | Baseline until the end of the study, up to approximately 9.5 months
  Number of participants with treatment emergent adverse events (TEAEs), serious adverse events (SAEs), and lab abnormalities according to NCI CTCAE Version 5.0
Part 1 and Part 2: Pharmacokinetic Parameter: Cmax of SAR443216 | From date of enrollment until the end of treatment, up to approximately 3.5 months for Part 1 and 5.5 months for Part 2
  Maximum observed plasma concentration
Part 1 and Part 2: Pharmacokinetic Parameter: Ctrough of SAR443216 | From date of enrollment until the end of treatment, up to approximately 3.5 months for Part 1 and 5.5 months for Part 2
  Plasma concentration observed just before treatment administration during repeated dosing
Part 1 and Part 2: Pharmacokinetic Parameter: t 1/2 of SAR443216 | From date of enrollment until the end of treatment, up to approximately 3.5 months for Part 1 and 5.5 months for Part 2
  Terminal half-life associated with the terminal slope (λz)
Part 1 and Part 2: Pharmacokinetic Parameter: AUC0-τ of SAR443216 | From date of enrollment until the end of treatment, up to approximately 3.5 months for Part 1 and 5.5 months for Part 2
  Area under the plasma concentration versus time curve
Part 1 and Part 2: Evaluation of SAR443216 immunogenicity | From date of enrollment until the end of treatment, up to approximately 3.5 months for Part 1 and 5.5 months for Part 2
  Incidence of ADA induction and ADA persistence

CONTACTS AND LOCATIONS:
Locations (11):
- ~University of Texas - MD Anderson Cancer Center Site Number : 8400002, Houston, Texas, United States
- Investigational Site Number : 0560002, Ghent, Belgium
- France (2):
  - Investigational Site Number : 2500001, Pierre-Bénite
  - Investigational Site Number : 2500002, Villejuif
- South Korea (2):
  - Investigational Site Number : 4100001, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100002, Seoul, Seoul-teukbyeolsi
- Spain (3):
  - Investigational Site Number : 7240003, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240001, Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7240002, Madrid / Madrid, Madrid, Comunidad de
- Taiwan (2):
  - Investigational Site Number : 1580001, Taichung
  - Investigational Site Number : 1580002, Tainan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: TED16925 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25361&tenant=MT_SNY_9011